CLINICAL TRIAL: NCT03741530
Title: Glibenclamide Advantage in Treating Edema After Intracerebral Hemorrhage (GATE-ICH): a Multi-center Randomized, Controlled, Assessor-blinded Trial
Brief Title: Glibenclamide Advantage in Treating Edema After Intracerebral Hemorrhage
Acronym: GATE-ICH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY20182067-X-3
Record Dates: First submitted 2018-11-08; First posted 2018-11-15 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2020-09

CONDITIONS: Intracerebral Hemorrhage
Keywords: Intracerebral hemorrhage; Perihematomal edema; Disability; Clinical trial
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — Glyburide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glibenclamide group (Experimental): Giving standard management for ICH plus glibenclamide tablets, 1.25 mg 3 times daily, orally or through gastric tube, for 7 consecutive days after enrollment.
  Interventions: Drug: Glibenclamide Tablets; Other: Standard management for ICH
- Control group (Placebo Comparator): Giving standard management for ICH
  Interventions: Other: Standard management for ICH

INTERVENTIONS:
Drug: Glibenclamide Tablets — Giving glibenclamide tablets, 1.25 mg 3 times daily, orally or through gastric tube, for 7 consecutive days after enrollment.
  Arms: Glibenclamide group
Other: Standard management for ICH — Usual care and drug in hospital

SUMMARY:
The purpose of the present study is to explore the efficacy of small doses of oral glibenclamide on brain edema after acute primary intracerebral hemorrhage (ICH), and improving the prognosis of patients.

DETAILED DESCRIPTION:
In order to explore the efficacy and safety of oral glibenclamide on brain edema after acute primary ICH, a web-based 1:1 randomization process will be employed to assign 220 subjects to Glibenclamide group (giving standard management for ICH plus glibenclamide) or Control group (giving standard management for ICH). The investigators will make a neurofunctional assessment at baseline, and 3 days, 7 days, 90 days after enrollment. The investigators also assess the midline shift, and the change in the volume of ICH and perihematomal edema (PHE) from the initial to follow-up (3 days and 7days after enrollment). The serious adverse events of all-cause mortality, cardiac-related and blood glucose-related adverse events will be collected to assess the safety of glibenclamide.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years with a primary ICH
2. A baseline CT with basal ganglia hemorrhage of 5 to 30 mL
3. Glasgow Coma Scale (GCS) score ≥ 6
4. Symptom onset less than 72 hours prior to admission
5. Informed consent

Exclusion Criteria:

1. Supratentorial ICH planned to evacuation of a large hematoma
2. Hemorrhage breaking into ventricles of brain
3. Prior significant disability (mRS ≥ 3)
4. Severe renal disease (i.e., renal disorder requiring dialysis ) or eGFR <30ml/min/1.73m2
5. Severe liver disorder, or ALT >3 times or bilirubin >2 times upper limit of normal
6. Blood glucose < 55 mg/dL (3.1 mmol/L）at enrollment, or with the history of hypoglycemia
7. With acute ST elevation infarction, or decompensated heart failure, or cardiac arrest, or acute coronary syndrome, or known history of admission for acute coronary syndrome, or acute myocardial infarction, or coronary intervention in the past 3 months
8. Treatment with sulfonylurea in the past 7 days, including glyburide, glyburide plus metformin, glimepiride, repaglinide, glipizide, gliclazide, tolbutamide and glibornuride
9. Treatment with bosentan in the past 7 days
10. Be allergic to sulfa or other sulfonylurea drugs
11. Known G6PD deficiency
12. Pregnant women
13. Breast-feeding women disagreeing to participate the study or stop breastfeeding during and after the study
14. Be enrolled in other non-observation-only study with receiving an investigational drug
15. Life expectancy <3 months due to other diseases rather than current ICH
16. Refusing to be enrolled, or having poor compliance, or tending to withdraw

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2020-09-23 (Actual); Study Completion 2020-09-23 (Actual)

PRIMARY OUTCOMES:
The proportion of death or major disability | 90 days after the onset
  Unfavourable outcome including death and disability is defined as patients achieving modified Rankin Scale (mRS) ≥3. The mRS is used for measuring the degree of disability or dependence in the daily activities of patients with stroke or other neurological diseases. The total score of the scale runs from 0 (perfect health without symptoms) to 6 (death).

SECONDARY OUTCOMES:
The change in the volume of ICH from the initial to follow-up CT scans | 3 days after onset
The change in the volume of PHE from the initial to follow-up CT scans | 3 days after onset
The change in the volume of ICH from the initial to follow-up CT scans | 7 days after onset
The change in the volume of PHE from the initial to follow-up CT scans | 7 days after onset
The proportion of death or major disability | 3 days after onset
  Unfavourable outcome including death and disability is defined as patients achieving modified Rankin Scale (mRS) ≥3. The mRS is used for measuring the degree of disability or dependence in the daily activities of patients with stroke or other neurological diseases. The total score of the scale runs from 0 (perfect health without symptoms) to 6 (death).
National Institute of Health stroke scale | 3 days after onset
  The National Institutes of Health Stroke Scale (NIHSS) is used by healthcare providers to evaluate the impairment caused by stroke. The total score of the scale runs from 0 to 42. The higher score is an indicative of more severe impairment.
Glasgow Coma Scale | 3 days after onset
  The Glasgow Coma Scale is a scale for measuring the conscious state of patients with neurological diseases. The total score of the scale runs from 3 (deep coma or death) to 15 (fully awake person).
Barthel Index | 3 days after onset
  The Barthel Index scale is used to measure performance in activities of daily living (ADL). The total score of the scale runs from 0 to 100. The high score of the scale represents favourable performance in activities of daily life.
The proportion of death or major disability | 7 days after onset
  Unfavourable outcome including death and disability is defined as patients achieving modified Rankin Scale (mRS) ≥3. The mRS is used for measuring the degree of disability or dependence in the daily activities of patients with stroke or other neurological diseases. The total score of the scale runs from 0 (perfect health without symptoms) to 6 (death).
National Institute of Health stroke scale | 7 days after onset
  The National Institutes of Health Stroke Scale (NIHSS) is used by healthcare providers to evaluate the impairment caused by stroke. The total score of the scale runs from 0 to 42. The higher score is an indicative of more severe impairment.
Glasgow Coma Scale | 7 days after onset
  The Glasgow Coma Scale is a scale for measuring the conscious state of patients with neurological diseases. The total score of the scale runs from 3 (deep coma or death) to 15 (fully awake person).
Barthel Index | 7 days after onset
  The Barthel Index scale is used to measure performance in activities of daily living (ADL). The total score of the scale runs from 0 to 100. The high score of the scale represents favourable performance in activities of daily life.
Barthel Index | 90 days after onset
  The Barthel Index scale is used to measure performance in activities of daily living (ADL). The total score of the scale runs from 0 to 100. The high score of the scale represents favourable performance in activities of daily life.

OTHER OUTCOMES:
Incidence of hypoglycemia | 7 days after admission
  Blood glucose <3.1 mmol/L
Incidence of symptomatic hypoglycemia | 7 days after admission
  Blood glucose <3.1 mmol/L with investigator-identified hypoglycemic symptoms
Incidence of cardiac-related Adverse Events and Serious Adverse Events | 7 days after admission
Incidence of all-cause mortality | 90 days after onset
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | During hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Wen Jiang, PhD, Study Director — Department of Neurology, Xijing Hospital, Fourth Military Medical
Locations (5):
- China (5):
  - Ankang Central Hospital, Ankang, Shaanxi
  - Hanzhong Central Hospital, Hanzhong, Shaanxi
  - Xijing Hospital, Xi'an, Shaanxi
  - Tangdu Hospital, Xi'an, Shaanxi
  - Xianyang Central Hospital, Xianyang, Shaanxi

REFERENCES:
- [Background] Keep RF, Hua Y, Xi G. Intracerebral haemorrhage: mechanisms of injury and therapeutic targets. Lancet Neurol. 2012 Aug;11(8):720-31. doi: 10.1016/S1474-4422(12)70104-7. Epub 2012 Jun 13. PMID 22698888
- [Background] Gebel JM Jr, Jauch EC, Brott TG, Khoury J, Sauerbeck L, Salisbury S, Spilker J, Tomsick TA, Duldner J, Broderick JP. Natural history of perihematomal edema in patients with hyperacute spontaneous intracerebral hemorrhage. Stroke. 2002 Nov;33(11):2631-5. doi: 10.1161/01.str.0000035284.12699.84. PMID 12411653
- [Background] Inaji M, Tomita H, Tone O, Tamaki M, Suzuki R, Ohno K. Chronological changes of perihematomal edema of human intracerebral hematoma. Acta Neurochir Suppl. 2003;86:445-8. doi: 10.1007/978-3-7091-0651-8_91. PMID 14753483
- [Background] Butcher KS, Baird T, MacGregor L, Desmond P, Tress B, Davis S. Perihematomal edema in primary intracerebral hemorrhage is plasma derived. Stroke. 2004 Aug;35(8):1879-85. doi: 10.1161/01.STR.0000131807.54742.1a. Epub 2004 Jun 3. PMID 15178826
- [Background] Xi G, Keep RF, Hoff JT. Mechanisms of brain injury after intracerebral haemorrhage. Lancet Neurol. 2006 Jan;5(1):53-63. doi: 10.1016/S1474-4422(05)70283-0. PMID 16361023
- [Background] Shi Y, Leak RK, Keep RF, Chen J. Translational Stroke Research on Blood-Brain Barrier Damage: Challenges, Perspectives, and Goals. Transl Stroke Res. 2016 Apr;7(2):89-92. doi: 10.1007/s12975-016-0447-9. Epub 2016 Jan 13. No abstract available. PMID 26757714
- [Background] Jiang B, Li L, Chen Q, Tao Y, Yang L, Zhang B, Zhang JH, Feng H, Chen Z, Tang J, Zhu G. Role of Glibenclamide in Brain Injury After Intracerebral Hemorrhage. Transl Stroke Res. 2017 Apr;8(2):183-193. doi: 10.1007/s12975-016-0506-2. Epub 2016 Nov 3. PMID 27807801
- [Derived] Zhao J, Song C, Li D, Yang X, Yu L, Wang K, Wu J, Wang X, Li D, Zhang B, Li B, Guo J, Feng W, Fu F, Gu X, Qian J, Li J, Yuan X, Liu Q, Chen J, Wang X, Liu Y, Wei D, Wang L, Shang L, Yang F, Jiang W; GATE-ICH Study Group. Efficacy and safety of glibenclamide therapy after intracerebral haemorrhage (GATE-ICH): A multicentre, prospective, randomised, controlled, open-label, blinded-endpoint, phase 2 clinical trial. EClinicalMedicine. 2022 Sep 23;53:101666. doi: 10.1016/j.eclinm.2022.101666. eCollection 2022 Nov. PMID 36177443
- [Derived] Zhao J, Yang F, Song C, Li L, Yang X, Wang X, Yu L, Guo J, Wang K, Fu F, Jiang W. Glibenclamide Advantage in Treating Edema After Intracerebral Hemorrhage (GATE-ICH): Study Protocol for a Multicenter Randomized, Controlled, Assessor-Blinded Trial. Front Neurol. 2021 Apr 27;12:656520. doi: 10.3389/fneur.2021.656520. eCollection 2021. PMID 33986719